CLINICAL TRIAL: NCT06608966
Title: Epilepsy Journey 2.0: An Intervention to Improve Executive Functioning in Adolescents With Epilepsy
Brief Title: Epilepsy Journey-An Executive Functioning Intervention for Teens With Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Medical University of South Carolina (Other); Children's Hospital of Orange County (Other); University of Georgia (Other); University of Iowa (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0297; UG3NS129558-01A1 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy in Children; Executive Dysfunction
Keywords: adolescents; executive functioning; seizures; epilepsy; behavioral trial; web-based intervention
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The proposed study will involve a multi-center randomized controlled clinical trial using a factorial design to simultaneously assess the impact of two behavioral treatment components: 1) Epilepsy Journey web-based modules and 2) Epilepsy Journey telehealth sessions with a therapist.There are four treatment arms for the current study, including 1) Epilepsy Journey web-based modules, 2) Epilepsy Journey web-based modules and telehealth with a therapist, 3) Telehealth with a therapist, and 4) Treatment as Usual.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI of the study is masked to treatment condition. Outcome assessors for the NIH toolbox measure will also be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Epilepsy Journey web-based modules alone (Experimental): Participants assigned to Epilepsy Journey modules will independently review web-based EJ modules. Participants will be targeted to complete 10 EJ modules (~15-30 minutes each session) within 14 weeks.
  Interventions: Behavioral: Epilepsy Journey web-based modules
- Epilepsy Journey web-based modules + telehealth with a therapist (Experimental): Participants will receive both the Epilepsy Journey web-based modules and telehealth sessions with a therapist weekly. Participants will review 10 modules independently (~15-30 minutes) and complete 10 telehealth sessions (~30-45 minutes each session) within a 14-week time frame.
  Interventions: Behavioral: Epilepsy Journey web-based modules; Behavioral: Telehealth with a therapist
- Telehealth with a therapist alone (Experimental): Participants will meet with a therapist for 10 telehealth sessions (30-45 minutes each session) within a 14-week time frame.
  Interventions: Behavioral: Telehealth with a therapist
- Treatment as Usual (No Intervention): Participants will receive no active behavioral health treatment components and will be followed in usual epilepsy care for 14 weeks.

INTERVENTIONS:
Behavioral: Epilepsy Journey web-based modules — Participants assigned to Epilepsy Journey modules will independently review web-based EJ modules focused on executive functioning skills. The modules cover 10 topic areas: Positive Thoughts, Problem-Solving, Initiation, Working Memory, Monitoring, Inhibition, Emotional Control, Organization and Planning, Sleep/Stress, and a Wrap-Up. Participants will complete 10 modules (~15-30 minutes each session) within a 14-week time frame. The goal is to complete one module per week.
  Arms: Epilepsy Journey web-based modules + telehealth with a therapist; Epilepsy Journey web-based modules alone
Behavioral: Telehealth with a therapist — Therapist will cover 10 areas of executive functioning during telehealth sessions, including Positive Thoughts, Problem-Solving, Initiation, Working Memory, Monitoring, Inhibition, Emotional Control, Organization and Planning, Sleep/Stress, and a Wrap-Up. Telehealth sessions with a therapist will occur via HIPAA-compliant videoconference (e.g. Microsoft Teams) each week ideally over the course of 14 weeks.
  Arms: Epilepsy Journey web-based modules + telehealth with a therapist; Telehealth with a therapist alone

SUMMARY:
The goal of this multi-site clinical trial is to determine the effectiveness of two components of a web-based intervention (Epilepsy Journey) to improve executive functioning in adolescents with epilepsy. The two components include web-based modules and problem-solving telehealth sessions with a therapist focused on executive functioning. This trial aims to answer the following questions:

1. Which components of Epilepsy Journey (web-based modules or telehealth sessions with a therapist) are essential for improving executive functioning in adolescents with epilepsy?
2. Which components of Epilepsy Journey (web-based modules or telehealth sessions with a therapist) are essential for improving quality of life in adolescents with epilepsy?

Participants will be randomly assigned to one of four groups: 1) Epilepsy Journey web-based modules and telehealth sessions, 2) Epilepsy Journey web-based modules only, 3) telehealth sessions with a therapist only, or 4) treatment as usual.

Participants will:

* Independently review Epilepsy Journey web-based modules focused on executive functioning skills (~15-30 minutes) and/or have weekly telehealth sessions (~30-45 minutes) with a therapist for 14 weeks.
* Complete measures of executive functioning (parent and teen-report) and quality of life (teen-report) at the start of the study, 14-, 26-, and 66- weeks after randomization. The NIH toolbox will be completed at the start of the study and 26-weeks after randomization. Additional measures will also be collected.

DETAILED DESCRIPTION:
Epilepsy is a common pediatric neurological condition affecting ~470,000 youth in the United States. Adolescents with epilepsy are at significant risk for neurobehavioral comorbidities (i.e., depressive/behavioral symptoms) and suboptimal social, academic, and quality of life outcomes. Research suggests that deficits in executive functioning (EF), defined as the skills necessary for goal-directed and complex activities, including problem-solving, initiation, monitoring, organization, planning, self-regulation and working memory, contribute to suboptimal functioning. EF deficits have been documented in up to 50% of youth with epilepsy, which is 3 times the prevalence in healthy youth. Evidence-based interventions to improve EF could play a critical role in preventing adverse outcomes and promoting optimal functioning in adolescents with epilepsy; however none exists for this vulnerable population. To fill this gap, the investigators successfully developed and tested Epilepsy Journey (EJ), a comprehensive e-health behavioral multi-component problem-solving intervention that combines 10 self-guided learning modules with 10 telehealth sessions. The promising proof-of-concept trial (n=39) showed high feasibility, acceptability, patient satisfaction, and significant improvements in parent-reported EF behaviors, neurobehavioral functioning, and quality of life. The next logical phase of this research is to conduct a definitive randomized clinical trial to examine: whether the two components of treatment (EJ modules and telehealth) are 1) both essential and 2) have a durable impact on improving parent-reported and performance-based EF behaviors and quality of life. Thus, the aim of the current proposal is to conduct a multi-site Phase 3 randomized controlled clinical trial (RCT) using a 2x2 factorial design to examine the efficacy of separate (EJ modules and EJ telehealth) and combined components of EJ on EF. Participants positive for EF deficits (n=232) will be randomized to one of four arms: 1) EJ modules with telehealth sessions, 2) EJ modules alone, 3) EJ telehealth sessions alone, or 4) Usual Care (no EJ modules or telehealth sessions). Treatment participants will either independently review EJ modules focused on EF skills (~15-30 min.) and/or have weekly telehealth sessions (~30-45 min.) with a therapist for 14-weeks. The groups will learn and apply problem-solving strategies to their individual EF difficulties. Participants will complete measures at baseline, 14-, 26-, and 66- weeks after randomization to examine maintenance of effects. There is a critical need for evidence-based interventions to improve executive functioning behaviors in youth with epilepsy. If the aims of this study are achieved, we will have definitive evidence for addressing EF deficits. The investigators expect that EJ modules and EJ telehealth will demonstrate efficacy alone and in combination, which will allow patients to select the approach best suited to their specific situation. Consequently, we can improve long-term outcomes (e.g., neurobehavioral comorbidities, academic success, social relationships, and quality of life) in adolescents with epilepsy, a high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 13-17 years at the time of enrollment
2. Child lives at home with primary caregiver and is enrolled in school (excluding summer breaks).
3. Confirmed diagnosis of epilepsy with seizures that are categorized as either generalized or focal in onset. Epilepsy is defined as: 1) At least two unprovoked seizures occurring more than 24-hours apart; or 2) One unprovoked seizure and a probability of further seizures similar to the general recurrence risk after two unprovoked seizures.
4. Primary language of English
5. Screening Inclusion: On the parent-reported Behavior Rating Inventory of Executive Function-2nd edition (BRIEF-2), have executive functioning deficits defined as at least 2 subclinical (60<T<65) or one clinical BRIEF-2 subscale T scores (T≥65).
6. Parent/legal guardian(s) willing to sign an IRB approved informed consent
7. Participant willing to sign an Institutional Review Board approved assent

Exclusion Criteria:

1. Parent or clinician-reported history in the adolescent of:

   1. developmental delay (e.g., autism spectrum disorder, pervasive development disorder, history of services for developmental delay or intellectual impairment in the past 5 years, known IQ<70)
   2. severe mental illness (e.g., schizophrenia, bipolar disorder, eating disorder within the past 12 months, depression with active suicidal ideation or suicidal ideation/intent in the past 3 months)
   3. prior (3-months) or current history of trauma and/or stressor-related disorders (e.g. PTSD)
   4. recent or current significant medical disease (i.e., cardiovascular, hepatic, renal, gynecologic, musculoskeletal, metabolic or endocrine)
   5. brain injury or brain tumor; and/or
   6. epilepsy surgery
   7. any other medical and/or psychological condition that takes treatment precedence over the study intervention
2. Clinician-reported diagnosis in the adolescent of

   1. epilepsy whose seizures are categorized only as either unknown onset or unclassified onset (defined as insufficient information to determine onset)
   2. epilepsy currently being treated at the time of enrollment by 3 or more antiseizure medications (ASMs) (excluding rescue medication use)
   3. epilepsy with a history of failure to achieve seizure freedom despite adequate use of 4 different anti-seizure medications
   4. a confirmed or suspected epileptic encephalopathy (e.g., electrical status epilepticus in sleep, Landau Kleffner syndrome, West syndrome)
   5. a confirmed or suspected progressive and degenerative disorder (e.g., mitochondrial disorders, metabolic disorders, autoimmune disorders)
   6. one or more episodes of status epilepticus within the 24 weeks prior to enrollment; and/or
   7. treatable causes of seizures, for example identified etiologies including metabolic, neoplastic, or active infectious origin.
   8. non-epileptic event/seizures
3. Adolescents currently on the ketogenic diet
4. Participation in a trial of an investigational drug or device within 30 days prior to screening

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function (2nd edition) Global Executive Composite T-score (parent) | 26-weeks post-randomization
  The parent-reported BRIEF-2 Global Executive Composite T-score will be used as the primary outcome measure. T-scores are linear transformations of raw scores, where 50 points represent the mean, and 10 points represent the standard deviation. T-scores provide information about an individual's score relative to a normal standardization sample, based on age and sex. T-scores ≥ 65 are considered clinically significant.

SECONDARY OUTCOMES:
PedsQL™ Epilepsy Module - Impact Subscale (Adolescent report) | 26-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific health-related quality of life (HRQOL) measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module - Cognitive Functioning Subscale (Adolescent report) | 26-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module - Executive Functioning Subscale (Adolescent report) | 26-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module -Sleep Subscale (Adolescent report) | 26-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module -Mood/Behavior Subscale (Adolescent report) | 26-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].

OTHER OUTCOMES:
Behavior Rating Inventory of Executive Function (2nd edition) -Global Executive Composite T-score (parent) | 66-weeks post-randomization
  The parent-reported BRIEF-2 GEC T-score will be used as the primary outcome measure. T-scores are linear transformations of raw scores, where 50 points represent the mean, and 10 points represent the standard deviation. T-scores provide information about an individual's score relative to a normal standardization sample, based on age and sex. T-scores ≥ 65 are considered clinically significant.
PedsQL™ Epilepsy Module - Impact Subscale (Adolescent report) | 66-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module - Cognitive Functioning Subscale (Adolescent report) | 66-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module - Executive Functioning Subscale (Adolescent report) | 66-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module -Sleep Subscale (Adolescent report) | 66-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
PedsQL™ Epilepsy Module -Mood/Behavior Subscale (Adolescent report) | 66-weeks post-randomization
  The PedsQL Epilepsy Module is reliable epilepsy-specific HRQOL measure for youth 2-25 years with epilepsy. Five key domains will be assessed, including Impact, Cognitive Functioning, Executive Functioning, Sleep, and Mood/Behavior. Scores range from 0-100, with higher scores representing better HRQOL. Clinical cut-offs have been established for the measure, with scores below the cut-off representing concerning HRQOL: Impact [Parent=60.7; Child=64.39], Cognitive [Parent=38.11; Child=50.97], Executive Functioning [Parent=46.65; Child=57.15], Sleep [Parent=42.07; Child=43.90], and Mood/Behavior [Parent=54.14; Child =53.30].
NIH Cognition Toolbox: Fluid Cognition Composite | 26-weeks post-randomization
  The Fluid Cognition Composite score will be calculated. Several subtests are included in the Fluid Cognition Composite, including Flanker (attention/inhibition), Dimensional Change Card Sorting (cognitive flexibility), Picture Sequent Memory (episodic memory); List Sorting (working memory); and Pattern Comparison (processing speed).
  A score at or near 100 indicates ability that is average compared with others nationally. Scores around 115 suggest above-average fluid cognitive ability, while scores around 130 suggest superior ability (in the top 2 percent nationally, based on Toolbox normative data). Conversely, a score around 85 suggests below-average fluid cognitive ability, and a score in the range of 70 or below suggests significant impairment, which may also be indicative of difficulties in school (for children) or general functioning.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Avani Modi, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Childrens Hospital of Orange County, Orange, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
This project will include demographic, medical, psychosocial and executive functioning data for adolescents with epilepsy. The raw questionnaire data and NIH Toolbox data will be stored within secure databases and environments. Protected Health Information (PHI) (e.g., respondent identifiers) will be restricted and maintained in a secure file until study results are published. All other scientific data (e.g., Scaled scores, contextual data) will be both preserved and shared. Prior to sharing, all data will be de-identified so that it is HIPAA-compliant.
  Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the NINDS Archived Clinical Research Datasets Repository, which houses NINDS clinical trial data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Final submission and release of the study data to the Archived Clinical Research Datasets Repository will occur at the time of publication of the primary manuscript or at the end of the performance period, whichever comes first. Study data deposited in the Repository will be available to the research community in perpetuity.
Access Criteria: All deidentified study data that are not designated as restricted use will be made available as public use data to the research community in accordance with the NINDS Archived Clinical Research Dataset Repository guidelines. Users of the public use data must register with NINDS and agree to the terms of use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting and prohibiting attempts to identify study participants. Data users also agree not to share or redistribute any data downloads. Further, users agree to destroy the dataset at the end of the research project.